CLINICAL TRIAL: NCT06801483
Title: Evaluation of the Effectiveness of Multiaxial Ankle Strengthening Training in Athletes With Chronic Ankle Instability
Brief Title: Ankle Strengthening in Athletes With Chronic Ankle Instability
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CMUH112-REC1-116(AR1); NSTC 113-2410-H-039-015 - (Other Grant/Funding Number: National Science and Technology Council, Taiwan)
Record Dates: First submitted 2025-01-21; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Chronic Ankle Instability, CAI; Athletes
Keywords: progressive training; strengthening; balance training; chronic ankle instability; ankle training machine
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multiaxial ankle training system (Experimental): These subjects will train their ankle strength by the multiaxial ankle training system
  Interventions: Other: Strengthening
- thera-band (Active Comparator): These subjects will train their ankle strength by thera-band
  Interventions: Other: Strengthening

INTERVENTIONS:
Other: Strengthening — All subjects will recieve an ankle muscle strenghening training program twice a week for six weeks.

SUMMARY:
Chronic ankle instability (CAI) is a common complication following an ankle sprain, affecting joint stability and leading to decreased muscle strength and poor neuromuscular control. These symptoms can significantly impact athletes' sports performance. Rehabilitation training for CAI majorly involves strengthening or balance training. Few studies have discussed treatment plans that combine the above two training, and the effectiveness of combined training is similar to that of single training content. Due to the lack of machines to train ankle strength, thera-bands were often used for ankle strengthening. However, the resistance thera-bands provide is limited and may need more for athletes requiring high-intensity training. In recent years, a local company has developed a multiaxial ankle training system for machine-based ankle strengthening. This machine allows for training the ankle joint in various directions while sitting and can provide greater training resistance. As this machine has recently been developed and there is seldom evidence for its use in training, this project aims to discuss the effectiveness of using the ankle training machine in athletes with chronic ankle instability. This study will compare the differences in muscle strength, morphology, muscle material properties, balance ability, and functional performance of athletes after a six-week combined training program with thera-band or the multiaxial ankle training system for providing resistance. Thereby establishing a training plan for athletes suffering from chronic ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral CAI: Cumberland Ankle Instability Tool (CAIT) score ≤ 24
* Age between 18 and 28 years
* Engages in sports training at least 3 days a week, for more than 1 hour each session
* Able to perform training and assessment movements

Exclusion Criteria:

* Bilateral CAI
* Less than 6 months since the first ankle sprain
* Acute ankle sprain within the last 6 weeks
* Foot or ankle surgery within the last 3 months
* Neuromuscular diseases.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Morphology | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  Using ultrasound to measure the muscle morphology of the peronous longus, gastrocnemius, tibialis anterior.
Y-Balance Test | At enrollment (1st week), midterm of training (3rd. week) and the end of training at 6 weeks
  This test is divided into three directions: anterior, posteromedial, and posterolateral. Each direction has a commercial measuring tape attached at 135 degrees, 90 degrees, and 135 degrees, respectively. The subject stands in the middle of the three measuring tapes, with the test foot's toe placed at the intersection point. The subject then stands on one leg with the test foot, extends the non-weight-bearing foot to touch the measuring tape in the target direction without touching the ground, and returns to the starting position while maintaining balance.
Countermovement Jump | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  Before the test, wireless EMG sensors are attached to the tibialis anterior, The test is performed on a force plate. The subject stands on the force plate, bends both knees to 90 degrees, and jumps as high as possible.
Triple Hop Test | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  The subject stands with both feet at the starting point in front of the force plate, then stands on one foot and performs three consecutive forward hops, with the first hop landing on the force plate.

SECONDARY OUTCOMES:
Ankle muscle strength | At enrollment (1st. week) and the end of intervention at 6 weeks
  Measuring muscle strength of dorsiflexion, plantarflexion, inversion and eversion by hand-hold dynamometer.
Muscle tension | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  The maximum values for muscle tension of tibialis anterior, lateral gastrocnemius, and peroneus longus muscles are evaluated by the MyotonPRO.
Muscle stiffness | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  The maximum values for muscle stiffness of tibialis anterior, lateral gastrocnemius, and peroneus longus muscles are evaluated by the MyotonPRO.
Muscle elasticity | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  The maximum values for muscle elasticity of tibialis anterior, lateral gastrocnemius, and peroneus longus muscles are evaluated by the MyotonPRO.
Muscle stress relaxation time | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  The maximum values for muscle stress relaxation time of tibialis anterior, lateral gastrocnemius, and peroneus longus muscles are evaluated by the MyotonPRO.
Muscle creep | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  The maximum values for muscle creep of tibialis anterior, lateral gastrocnemius, and peroneus longus muscles are evaluated by the MyotonPRO.
Eyes Open/Eyes Closed Single-Leg Stance Test | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  This test includes static single-leg stance with eyes open/closed on stable/unstable surfaces, using a force plate to record the center of pressure changes during the test. The starting posture is single-leg stance with hands on hips and the non-test foot lightly touching the inner ankle of the weight-bearing foot. The subject maintains stable standing for 30 seconds. If instability occurs, hands and feet can leave the body to maintain balance, but the test foot must not move. If the other foot touches the ground, the test is considered a failure. For the unstable surface test, a soft pad is placed on the force plate, and the subject stands on the pad.
Muscle activation during countermovement Jump | At enrollment (1st. week), midterm of training (3rd. week) and the end of training at 6 weeks
  The wireless EMG sensors are attached to the tibialis anterior, peroneus longus, and lateral gastrocnemius muscles to capture muscle activation during the activity.
Foot and Ankle Ability Measure (FAAM) | At enrollment (1st. week) and the end of training at 6 weeks
  The Foot and Ankle Ability Measure (FAAM) is a self-reported functional assessment for the ankle joint, divided into two domains: Activities of Daily Living (FAAM-ADL) and Sports (FAAM-Sports), with 21 and 8 items, respectively. Subjects rate the difficulty of performing each activity based on their perception, with 4 points for no difficulty and 0 points for unable to perform.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ming Chang, Ph.D., Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No